CLINICAL TRIAL: NCT06006585
Title: Safety, Tolerability, and Pharmacokinetics of Intravitreal Single Rising Doses and Multiple Doses of BI 771716 in Patients With Geographic Atrophy Secondary to Age-related Macular Degeneration (Open Label, Non-randomized)
Brief Title: A Study to Test How Well Different Doses of BI 771716 Are Tolerated by People With an Advanced Form of Age-related Macular Degeneration (AMD) Called Geographic Atrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1497-0001
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 771716 low dose treatment group (Single rising dose (SRD part)) (Experimental)
  Interventions: Drug: BI 771716
- BI 771716 treatment group (multiple dose (MD part)) (Experimental)
  Interventions: Drug: BI 771716
- BI 771716 medium dose treatment group (SRD part) (Experimental)
  Interventions: Drug: BI 771716
- BI 771716 high dose treatment group (SRD part) (Experimental)
  Interventions: Drug: BI 771716

INTERVENTIONS:
Drug: BI 771716 — BI 771716

SUMMARY:
This study is open to adults with geographic atrophy, an advanced form of age-related macular degeneration. People can join the study if they are at least 50 years old. The purpose of this study is to find out how well different doses of a medicine called BI 771716 are tolerated.

This study has 2 parts. Part 1 of the study takes about 3 months. In this part, participants receive 1 injection of BI 771716 directly into one of the eyes affected by geographic atrophy.

Part 2 of the study takes about 4 months. In this part, participants receive 2 injections of BI 771716 directly into the eye. There are 4 weeks between the first and the second injection. In this study, BI 771716 is given to humans for the first time.

The doctors compare how well participants tolerate the different doses of BI 771716. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with geographic atrophy (GA) secondary to age-related macular degeneration (AMD), with any GA lesion of minimum 1 disc diameter (minimum 2.5 mm^2) in size, and unlimited maximum size. This may include GA lesions contiguous to or continuous with peripapillary atrophy.
2. Fellow eye is not required to have GA.
3. Best corrected visual acuity (BCVA) in the non-study eye must have a better BCVA compared to the study eye.
4. BCVA of ≥4 and ≤70 letters in the study eye (approximate equivalent to 20/800 and 20/40 on the Snellen chart) measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol.
5. Age at least 50 years.
6. Men able to father a child must be ready and able to use highly effective methods of birth control per the International Council on Harmonisation of Technical Requirements for Registration of Human Use guideline M3(R2) (ICH M3(R2)) that would result in a low failure rate of less than 1% per year when used consistently and correctly.
7. Signed informed consent consistent with ICH good clinical practice (GCP) guidelines and local legislation prior to participation in the trial, which includes medication washout and restrictions.
8. Not under any administrative or legal supervision or under institutionalization due to regulatory or juridical order.

Exclusion Criteria:

1. Women of childbearing potential (WOCBP) cannot be included. A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy or another cause as determined by the investigator (e.g. Müllerian agenesis). Tubal ligation is NOT a method of permanent sterilization. A postmenopausal state is defined as no menses for 1 year without an alternative medical cause.
2. History of or evidence of current active exudative choroidal neovascularization (CNV) in the study eye. History of evidence of exudative CNV in the fellow eye is not exclusionary. Eyes with evidence of non-exudative CNV are not exclusionary (as identified by spectral domain optical coherence tomography (SD-OCT) and fluorescein angiography (FA)) .
3. Previously received treatment in the study eye for GA secondary to AMD within 3 months prior to screening.
4. Previous trial participation receiving trial medication for GA in the study eye secondary to AMD within 6 months prior to screening. Use of any investigational drug within 90 days or 5 half-lives prior to screening, whichever is longer.
5. Previously received gene therapy or cell therapy.
6. Additional eye disease in the study eye that could compromise trial participation:

   1. uncontrolled glaucoma or intraocular pressure >24 mmHg.
   2. clinically significant diabetic maculopathy.
   3. history of high myopia >8 diopters in the study eye.
   4. anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation with Spectral domain optical coherence tomography (SD-OCT).
   5. exclude ocular conditions at discretion of the investigator that might interfere with outcome of the trial.
7. Exclude prior vitrectomy surgery.
8. Exclude study eyes that have undergone glaucoma drainage implantation or trabeculectomy. History of microinvasive glaucoma surgery may be included.

Further exclusion criteria apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Occurrence of ocular dose limiting events (DLEs) from drug administration until Day 8 | Up to 7 days
  SRD part
Occurrence of drug-related adverse events (AEs) from drug administration until end of study (EOS) | Up to 112 days
  MD part

SECONDARY OUTCOMES:
Occurrence of any ocular adverse events (AEs) in the study eye from drug administration until EOS | Up to 112 days
  SRD part
Maximum serum concentration of BI 771716 after a single intravitreal (IVT) dose (Cmax) | Up to 84 days
  SRD part
Area under the concentration-time curve of BI 771716 in serum over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 84 days
  SRD part
Time from dosing to maximum serum concentration of BI 771716 (tmax) | Up to 84 days
  SRD part
Trough concentration of BI 771716 in serum | At Day 29
  MD part
BI 771716 serum concentration | At Day 57
  MD part

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Bay Area Retina Associates - Walnut Creek, Walnut Creek, California
  - Florida Retina Institute, Jacksonville, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Verum Research, LLC, Eugene, Oregon
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Tennessee Retina, Nashville, Tennessee
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Houston, PA-Houston-62050, Houston, Texas
  - Retina Consultants of Texas-The Woodlands-67575, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com